CLINICAL TRIAL: NCT00670644
Title: Breast Cancer Treatment Related Lymphedema Self Care Practices
Brief Title: Self-Care for Lymphedema in Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sheila Ridner, Professor, Vanderbilt University
Other Study IDs: CDR0000587714; P30CA068485 (NIH); VU-VICC-SUPP-0628; VU-VICC-060480
Record Dates: First submitted 2008-05-01; First posted 2008-05-02 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: questionnaire administration — Completed self-report form
Other: survey administration — Completed self-report form-other
Procedure: quality-of-life assessment — Completed self-report form qol

SUMMARY:
RATIONALE: Identifying why patients don't do self care for lymphedema may help doctors plan better at-home self-care treatment.

PURPOSE: This research study is looking at self-care practices for lymphedema in patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To systematically identify and describe the barriers to completing recommended at home self-care of lymphedema in patients with breast cancer.
* To identify patient recalled instructions as to at home self-care practices for lymphedema as told to them by healthcare professionals and others.
* To identify the current at home self-care practices of breast cancer survivors with treatment treated lymphedema.

Secondary

* To examine the relationship between at home self-care activities and symptoms in breast cancer survivors with lymphedema.
* To examine the relationship between at home self-care activities and quality of life in breast cancer survivors with lymphedema.
* To identify patient-perceived benefits to at home self-care.

OUTLINE: Patients complete questionnaires about their breast cancer diagnosis and treatment history, lymphedema history and problems, and years of education and income. Patients also complete surveys about home self-care practices for lymphedema and any benefits, burdens, or barriers of at home care.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of breast cancer
* Lymphedema in one or both arms that occurred during or after breast cancer treatment
* Must have received prior lymphedema treatment by a healthcare professional

  * Patients with self-reported arm swelling subsequent to breast cancer treatment that has not been treated by a healthcare professional are not eligible
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* English speaking

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Identification and description of barriers to completing recommended at home self-care of lymphedema | one time only for approximately 15 minutes
Identification of patients recalled instructions as to at home self-care practices for lymphedema as told to them by healthcare professionals and others | one time only for approximately 15 minutes
Identification of current at home self-care practices for lymphedema | one time only for approximately 15 minutes

SECONDARY OUTCOMES:
Relationship between at home self-care activities, symptoms, and quality of life in breast cancer survivors with lymphedema | one time only for approximately 15 minutes
Identification of patient-perceived benefits to at home self-care | one time only for approximately 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Shiela H. Ridner, MSN, PhD, RN, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee